CLINICAL TRIAL: NCT01083186
Title: Paricalcitol Oral Therapy in Predialysis CKD Patients. The Greek Experience
Acronym: PROTECT
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P11-978
Record Dates: First submitted 2010-02-20; First posted 2010-03-09 (Estimated); Results first posted 2013-03-07 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Kidney Failure; Secondary Hyperparathyroidism
Keywords: Secondary Hyperparathyroidism; Chronic Kidney Failure
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperparathyroidism, Secondary

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism: Participants with chronic kidney disease stage 3-5 with secondary hyperparathyroidism, who were prescribed oral paricalcitol according to the approved Summary of Product Characteristics (SmPC)

SUMMARY:
The purpose of this study is to obtain data on the use of Zemplar (paricalcitol) capsules in real-life clinical practice in predialysis patients with chronic kidney disease (CKD) and secondary hyperparathyroidism.

DETAILED DESCRIPTION:
This was a single arm, open, multicenter, non-interventional, post marketing observational study, which has been conducted in 24 sites in Greece, under normal clinical practice and as per the locally approved Summary of Product Characteristics (SmPC) of study medication (oral paricalcitol). Eligible patients were followed up for a 12-month period after enrollment. All study activities were consistent with European Union (EU) directive 2001/20/EC section for non-interventional studies.

In this study, paricalcitol was prescribed on an on-label basis in an everyday setting to observe drug actions in a distinct geography (Greece with > 250 days/year of sunny days) as well as in a significant subpopulation (Chronic Kidney Disease [CKD] stages 3-5 transplanted patients). Dose tolerability, treatment effects, as well as maintenance of results were registered for a 12-month period in order to obtain experience in the long term use of paricalcitol capsules. Furthermore, in centers where additional blood parameters were examined as part of clinical routine, these were recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with secondary hyperparathyroidism in the presence of chronic kidney disease stage 3, 4 or 5 treated with Zemplar (paricalcitol) oral for at least 1 month prior to study enrollment
* Male and female (not pregnant or not planning to be pregnant in the next 12 months) patients > 18 years of age
* Signed informed consent by subject
* Hypertensive and diabetic subjects must be on an optimal and steady medication regimen for more than 30 days

Exclusion Criteria:

* Contraindications listed in the Summary of Product Characteristics for Zemplar capsules apply (Appendix I and II)
* Parathormone value of > 1000 pg/mL (sign of tertiary hyperparathyroidism)
* Treatment with Vitamin D within the last 1 month prior to inclusion into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from 24 hospital-based specialty, nephrology clinics in Greece
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Argyropoulos, MD, Study Director — AbbVie Pharmaceuticals S.A.
Locations (24):
- Greece (24):
  - Site Reference ID/Investigator# 47002, Arta
  - Site Reference ID/Investigator# 43772, Athens
  - Site Reference ID/Investigator# 27492, Athens
  - Site Reference ID/Investigator# 43769, Athens
  - Site Reference ID/Investigator# 38257, Athens
  - Site Reference ID/Investigator# 47003, Athens
  - Site Reference ID/Investigator# 27497, Athens
  - Site Reference ID/Investigator# 47004, Athens
  - Site Reference ID/Investigator# 27489, Athens
  - Site Reference ID/Investigator# 27495, Athens
  - Site Reference ID/Investigator# 43773, Athens
  - Site Reference ID/Investigator# 27498, Haidari, Athens
  - Site Reference ID/Investigator# 38259, Ioannina
  - Site Reference ID/Investigator# 22121, Larissa
  - Site Reference ID/Investigator# 43771, Larissa
  - Site Reference ID/Investigator# 43767, Maroussi Athens
  - Site Reference ID/Investigator# 27496, Nikaia
  - Site Reference ID/Investigator# 43768, North Ionia, Athens
  - Site Reference ID/Investigator# 27491, Piraeus
  - Site Reference ID/Investigator# 27494, Thessaloniki
  - Site Reference ID/Investigator# 27493, Thessaloniki
  - Site Reference ID/Investigator# 38255, Thessaloniki
  - Site Reference ID/Investigator# 43770, Thessaloniki
  - Site Reference ID/Investigator# 39839, Thessaloniki

REFERENCES:
- See also: Related info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Started | 500
Completed | 406
Not Completed | 94
Not completed — Lost to Follow-up | 48
Not completed — Consent Withdrawal | 7
Not completed — Death | 3
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 2
Not completed — Hemodialysis Initiation | 28
Not completed — Administrative Reasons | 2
Not completed — Non-compliance to Study Treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
Age Continuous [Mean (Standard Deviation); unit: years] | 67.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186
  Male | 314

OUTCOME MEASURES:

1. Primary Outcome: Intact Parathormone (iPTH) Changes During the Study Time-Points for Overall Study Population
Description: iPTH levels before and after oral paricalcitol treatment onset were recorded at each study visit, and corresponding changes were calculated for the overall study population.
Time Frame: Baseline, Enrollment Visit, Month 3, Month 6, Month 9, Month 12
Population: Overall study population. n=number of participants with available data at given time-point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
pg/mL
  Before Study Treatment (Baseline); n=495 | 232.1 (168.2)
  Visit 1 (Enrollment); n=497 | 200.1 (141.1)
  Visit 2 (3 Months Post-Enrollment); n=432 | 166.6 (137.6)
  Visit 3 (6 Months Post-Enrollment); n=405 | 157.3 (172.9)
  Visit 4 (9 Months Post-Enrollment); n=378 | 135.2 (99.5)
  Visit 5 (12 Months Post-Enrollment); n=368 | 119.4 (63.1)
  Change from Baseline to Enrollment; n=492 | -32.2 (96.0)
  Change from Baseline to Visit 2; n=429 | -62.6 (125.5)
  Change from Baseline to Visit 3; n=402 | -69.7 (172.4)
  Change from Baseline to Visit 4; n=376 | -85.4 (129.4)
  Change from Baseline to Visit 5; n=364 | -96.1 (130.8)
  Change from Enrollment to Visit 2; n=430 | -35.6 (93.2)
  Change from Enrollment to Visit 3; n=404 | -41.9 (150.4)
  Change from Enrollment to Visit 4; n=378 | -58.4 (112.4)
  Change from Enrollment to Visit 5; n=367 | -72.4 (113.4)

2. Primary Outcome: Intact Parathormone (iPTH) Changes During the Study Time-Points for Subpopulation of Renal Transplanted Participants
Description: iPTH levels before and after oral paricalcitol treatment onset were recorded at each study visit, and corresponding changes were calculated for the subpopulation of renal transplanted participants.
Time Frame: Baseline, Enrollment Visit, Month 3, Month 6, Month 9, Month 12
Population: Participants with renal transplantation history. n=number of participants with available data at given time-point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 40
pg/mL
  Before Study Treatment (Baseline); n=40 | 321.5 (293.6)
  Visit 1 (Enrollment); n=39 | 269.3 (214.5)
  Visit 2 (3 Months Post-Enrollment); n=27 | 240.1 (166.0)
  Visit 3 (6 Months Post-Enrollment); n=21 | 271.4 (225.2)
  Visit 4 (9 Months Post-Enrollment); n=15 | 299.7 (231.9)
  Visit 5 (12 Months Post-Enrollment); n=21 | 182.9 (109.6)
  Change from Baseline to Enrollment; n=39 | -50.1 (144.8)
  Change from Baseline to Visit 2; n=27 | -93.0 (134.8)
  Change from Baseline to Visit 3; n=21 | -95.4 (262.0)
  Change from Baseline to Visit 4; n=15 | -71.3 (228.2)
  Change from Baseline to Visit 5; n=21 | -92.5 (139.4)
  Change from Enrollment to Visit 2; n=26 | -61.3 (106.1)
  Change from Enrollment to Visit 3; n=20 | -72.1 (215.0)
  Change from Enrollment to Visit 4; n=15 | -69.0 (207.3)
  Change from Enrollment to Visit 5; n=20 | -73.1 (144.6)

3. Secondary Outcome: Median Time to Attain the First Lower Intact Parathormone (iPTH) Levels
Description: The time to attain the first lower iPTH levels was considered as the time from the date of oral paricalcitol treatment onset until the date when any of the following conditions were initially met: a 30% reduction from iPTH levels prior to treatment onset had been achieved, for patients who were still outside the target range; or iPTH levels equal or lower to the upper limit of the target range according to Kidney Disease Quality Outcome Initiative (K/DOQI) guidelines (CKD Stage 3: ≤ 70 pg/mL; CKD Stage 4: ≤ 110 pg/mL; CKD Stage 5: ≤ 300 pg/mL).
Time Frame: Measured from start of study, up to a maximum of 12 months
Population: Subset of participants with baseline CKD stage ≥ 3 as well as with available iPTH values greater than the upper limit of the target range, prior to paricalcitol treatment onset. Target range for this specific analysis was defined based on patient's CKD stage (per baseline eGFR) prior to paricalcitol treatment onset.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 470
months | 7.8 [7.2 to 8.5]

4. Secondary Outcome: Mean Duration of Effect Sustainability (Months)
Description: The effect was considered sustainable if: the participant's intact parathormone (iPTH) value remained equal or lower to the upper limit of the target range according to Kidney Disease Quality Outcome Initiative (K/DOQI) guidelines (CKD Stage 3: ≤ 70 pg/mL; CKD Stage 4: ≤ 110 pg/mL); or iPTH levels continued to decrease 30% from the previous available measurement.
Time Frame: Measured from start of study, up to a maximum of 12 months
Population: All evaluable participants
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 362
months | 3.8 (2.4)

5. Secondary Outcome: Distribution of Participants by Achievement of Intact Parathormone (iPTH) Levels Within the Target Range
Description: Number of participants with iPTH levels within the target range of Kidney Disease Quality Outcome Initiative (K/DOQI) treatment guidelines at each study measurement after oral paricalcitol treatment onset. K/DOQI treatment guidelines: CKD Stage 3: 35-70 pg/mL; CKD Stage 4: 70-110 pg/mL during a 12-month period of treatment with oral paricalcitol.
Time Frame: Enrollment Visit, Month 3, Month 6, Month 9, Month 12
Population: All participants. n=participants with evaluable data at given time point.
Measure: Number; unit: participants
Groups:
- Participants Within the iPTH Target Range: Number of participants with iPTH levels within the target range of K/DOQI treatment guidelines: CKD Stage 3: 35-70 pg/mL; CKD Stage 4: 70-110 pg/mL during a 12-month period of treatment with oral paricalcitol.
- Participants Out of the iPTH Target Range: Number of participants with iPTH levels outside of the target range of K/DOQI treatment guidelines: CKD Stage 3: 35-70 pg/mL; CKD Stage 4: 70-110 pg/mL during a 12-month period of treatment with oral paricalcitol.
Arm/Group | Participants Within the iPTH Target Range | Participants Out of the iPTH Target Range
Number analyzed (Participants) | 500 | 500
participants
  Visit 1 (Enrollment); n=497 | 11 | 486
  Visit 2 (3 Months Post-Enrollment); n=432 | 75 | 357
  Visit 3 (6 Months Post-Enrollment); n=405 | 76 | 329
  Visit 4 (9 Months Post-Enrollment); n=378 | 89 | 289
  Visit 5 (12 Months Post-Enrollment); n=368 | 101 | 267

6. Secondary Outcome: Number of Participants With Serum Calcium Level Abnormalities
Description: Normal serum calcium range was 8.4-10.2 mg/dL.
Time Frame: Baseline, Enrollment Visit, Month 6, Month 12
Population: All participants. n=number of participants with evaluable data at given time-point.
Measure: Number; unit: participants
Groups:
- Participants Within the Normal Calcium Range; Participants Outside of the Normal Calcium Range: Normal serum calcium range was 8.4-10.2 mg/dL.
Arm/Group | Participants Within the Normal Calcium Range | Participants Outside of the Normal Calcium Range
Number analyzed (Participants) | 500 | 500
participants
  Before Study Treatment (Baseline); n=461 | 384 | 77
  Visit 1 (Enrollment); n=471 | 409 | 62
  Visit 3 (6 Months Post-Enrollment); n=436 | 391 | 45
  Visit 5 (12 Months Post-Enrollment); n=386 | 342 | 44

7. Secondary Outcome: Number of Participants With Serum Phosphorus Level Abnormalities
Description: Normal serum phosphorus range was 2.7-4.6 mg/dL.
Time Frame: Baseline, Enrollment Visit, Month 6, Month 12
Population: All participants. n=number of participants with evaluable data at given time-point
Measure: Number; unit: participants
Groups:
- Participants Within the Phosphorus Normal Range; Participants Outside of the Phosphorus Normal Range: Normal serum phosphorus range was 2.7-4.6 mg/dL.
Arm/Group | Participants Within the Phosphorus Normal Range | Participants Outside of the Phosphorus Normal Range
Number analyzed (Participants) | 500 | 500
participants
  Before Study Treatment (Baseline); n=451 | 367 | 84
  Visit 1 (Enrollment); n=466 | 361 | 105
  Visit 3 (6 Months Post-Enrollment); n=429 | 326 | 103
  Visit 5 (12 Months Post-Enrollment); n=375 | 271 | 104

8. Secondary Outcome: Change in Dipstick Albuminuria Grade From Baseline to Month 6
Description: The values "-, Trace, +, ++, and +++" are taken directly from the dipstick measurements, and represent a range from none to highest albuminuria. Data presented shows the number of participants with each value both at Baseline and at Month 6.
Time Frame: Baseline, Month 6
Population: Number of participants with evaluable data at both Baseline and Visit 3 (6 Months Post-Enrollment)
Measure: Number; unit: participants
Groups:
- No Albuminuria at Month 6: The value "-" is taken directly from the dipstick measurements, and represents a reading of no albuminuria.
- Trace Albuminuria at Month 6: The value "Trace" is taken directly from the dipstick measurements, and represents a reading of trace albuminuria.
- "+" Albuminuria at Month 6: The value "+" is taken directly from the dipstick measurements, and represents the middle of a range from none to highest albuminuria.
- "++" Albuminuria at Month 6: The value "++" is taken directly from the dipstick measurements, and represents the value second to highest albuminuria.
- "+++" Albuminuria at Month 6: The value "+++" is taken directly from the dipstick measurements, and represents the highest albuminuria.
Arm/Group | No Albuminuria at Month 6 | Trace Albuminuria at Month 6 | "+" Albuminuria at Month 6 | "++" Albuminuria at Month 6 | "+++" Albuminuria at Month 6
Number analyzed (Participants) | 162 | 162 | 162 | 162 | 162
participants
  Grade "-" at Baseline | 19 | 1 | 10 | 2 | 0
  Grade "Trace" at Baseline | 1 | 0 | 1 | 0 | 0
  Grade "+" at Baseline | 15 | 1 | 36 | 10 | 3
  Grade "++" at Baseline | 2 | 0 | 9 | 18 | 4
  Grade "+++" at Baseline | 0 | 2 | 7 | 6 | 15

9. Secondary Outcome: Change in Dipstick Albuminuria Grade From Baseline to Month 12
Description: as for outcome 8
Time Frame: Baseline, Month 12
Population: Number of participants with evaluable data at both Baseline and Visit 5 (12 Months Post-Enrollment)
Measure: Number; unit: participants
Groups:
- No Albuminuria at Month 12: The value "-" is taken directly from the dipstick measurements, and represents a reading of no albuminuria.
- Trace Albuminuria at Month 12: The value "Trace" is taken directly from the dipstick measurements, and represents a reading of trace albuminuria.
- "+" Albuminuria at Month 12: The value "+" is taken directly from the dipstick measurements, and represents the middle of a range from none to highest albuminuria.
- "++" Albuminuria at Month 12: The value "++" is taken directly from the dipstick measurements, and represents the value second to highest albuminuria.
- "+++" Albuminuria at Month 12: The value "+++" is taken directly from the dipstick measurements, and represents the highest albuminuria.
Arm/Group | No Albuminuria at Month 12 | Trace Albuminuria at Month 12 | "+" Albuminuria at Month 12 | "++" Albuminuria at Month 12 | "+++" Albuminuria at Month 12
Number analyzed (Participants) | 149 | 149 | 149 | 149 | 149
participants
  Grade "-" at Baseline | 18 | 3 | 6 | 3 | 0
  Grade "Trace" at Baseline | 0 | 0 | 1 | 0 | 0
  Grade "+" at Baseline | 14 | 1 | 37 | 9 | 2
  Grade "++" at Baseline | 2 | 0 | 8 | 13 | 5
  Grade "+++" at Baseline | 0 | 0 | 6 | 1 | 20

10. Secondary Outcome: Glycosylated Hemoglobin A1c (HbA1c) Values Throughout the Study
Description: The HbA1c normal range was 4.3-6.1%.
Time Frame: Baseline, Enrollment Visit, Month 6, Month 12
Population: All participants. n=number of participants with evaluable data at given time-points.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
percent
  Before Study Treatment (Baseline); n=101 | 7.2 (1.6)
  Visit 1 (Enrollment); n=99 | 6.9 (1.4)
  Visit 3 (6 Months Post-Enrollment); n=76 | 7.0 (1.5)
  Visit 5 (12 Months Post-Enrollment); n=69 | 6.9 (1.2)

11. Secondary Outcome: Non-serious Adverse Events (nSAEs) and Serious Adverse Events (SAEs)
Description: In order to establish the safety profile of oral paricalcitol in daily clinical practice, non-serious adverse events (nSAEs) and serious adverse events (SAEs) were collected during the course of the study. An adverse event (AE) is defined as any untoward medical occurrence in a patient, which does not necessarily have a causal relationship with their treatment. If an adverse event meets any of the following criteria, it is considered a serious adverse event (SAE): results in death or is life-threatening, results in admission or prolongation of hospitalization, is a congenital anomaly or persistent or significant disability/incapacity or is an important medical event requiring medical or surgical intervention to prevent any of the outcomes listed above. Please see Adverse Events section below for more details.
Time Frame: From time of enrollment throughout the study up to 12 months for nSAEs. SAEs from time of enrollment throughout the study up to + 30 days after end of study.
Population: All participants
Measure: Number; unit: participants
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
participants
  Adverse Events (nSAEs and SAEs) | 192
  nSAEs | 180
  SAEs | 19

12. Secondary Outcome: Distribution of Participants by Chronic Kidney Disease (CKD) Stage Throughout Study
Description: Change in CKD stage throughout the study period was assessed by the estimated glomerular filtration rate (eGFR) levels recorded by the physicians at each study time point. Classification of eGFR into CKD stages as follows: CKD stage 2: 60-89 mL/min/1.73m^2; CKD stage 3: 30-59 mL/min/1.73m^2; CKD stage 4: 15-29 mL/min/1.73m^2; CKD stage 5: <15 mL/min/1.73/m^2. Table presents the number of participants by stage at each study visit.
Time Frame: Baseline, Enrollment Visit, Month 3, Month 6, Month 9, Month 12
Population: All participants. n=number of participants with evaluable data at given time-points.
Measure: Number; unit: participants
Groups:
- CKD Stage 2: Participants with chronic kidney disease stage 2 (eGFR 60-89 mL/min/1.73m^2) with secondary hyperparathyroidism, who were prescribed oral paricalcitol according to the approved Summary of Product Characteristics (SmPC)
- CKD Stage 3: Participants with chronic kidney disease stage 3 (eGFR 30-59 mL/min/1.73m^2)with secondary hyperparathyroidism, who were prescribed oral paricalcitol according to the approved Summary of Product Characteristics (SmPC)
- CKD Stage 4: Participants with chronic kidney disease stage 4 (eGFR 15-29 mL/min/1.73m^2)with secondary hyperparathyroidism, who were prescribed oral paricalcitol according to the approved Summary of Product Characteristics (SmPC)
- CKD Stage 5: Participants with chronic kidney disease stage 5 (eGFR <15 mL/min/1.73m^2)with secondary hyperparathyroidism, who were prescribed oral paricalcitol according to the approved Summary of Product Characteristics (SmPC)
Arm/Group | CKD Stage 2 | CKD Stage 3 | CKD Stage 4 | CKD Stage 5
Number analyzed (Participants) | 500 | 500 | 500 | 500
participants
  Visit 1 (Enrollment); n=500 | 0 | 234 | 266 | 0
  Visit 2 (3 Months Post-Enrollment); n=463 | 2 | 214 | 214 | 33
  Visit 3 (6 Months Post-Enrollment); n=451 | 3 | 197 | 210 | 41
  Visit 4 (9 Months Post-Enrollment); n=426 | 3 | 190 | 185 | 48
  Visit 5 (12 Months Post-Enrollment); n=406 | 1 | 175 | 184 | 46

13. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) Values Throughout the Study
Description: The eGFR normal range was 90-120 mL/min/1.73m^2.
Time Frame: Baseline, Enrollment Visit, Month 3, Month 6, Month 9, Month 12
Population: All participants. n=number of participants with evaluable data at given time-points.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
mL/min/1.73m^2
  Before Study Treatment (Baseline); n=499 | 30.4 (11.3)
  Visit 1 (Enrollment); n=500 | 29.9 (11.3)
  Visit 2 (3 Months Post-Enrollment); n=463 | 29.6 (12.2)
  Visit 3 (6 Months Post-Enrollment); n=451 | 29.6 (12.4)
  Visit 4 (9 Months Post-Enrollment); n=426 | 29.6 (12.6)
  Visit 5 (12 Months Post-Enrollment); n=406 | 29.1 (12.4)

14. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT) Levels at Months 6 and 12
Description: The alanine aminotransferase normal range was 11-43 IU/L.
Time Frame: Baseline, Month 6, Month 12
Population: All participants. n=number of participants with evaluable data at given time-points.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
IU/L
  Before Study Treatment (Baseline); n=367 | 20.2 (10.2)
  Change from Baseline to Visit 3 (6 Months); n=276 | -0.4 (11.0)
  Change from Baseline to Visit 5 (12 months); n=259 | 0.3 (11.3)

15. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) Levels at Months 6 and 12
Description: The aspartate aminotransferase normal range was 11-38 IU/L.
Time Frame: Baseline, Month 6, Month 12
Population: All participants. n=number of participants with evaluable data at given time-points.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
IU/L
  Before Study Treatment (Baseline); n=365 | 21.1 (10.3)
  Change from Baseline to Visit 3 (6 Months); n=276 | 0.0 (10.6)
  Change from Baseline to Visit 5 (12 months); n=257 | -0.9 (10.8)

16. Secondary Outcome: Change From Baseline in Creatinine Levels at Months 6 and 12
Description: The creatinine normal range was 0.6-1.4 mg/dL.
Time Frame: Baseline, Month 6, Month 12
Population: All participants. n=number of participants with evaluable data at given time-points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
mg/dL
  Before Study Treatment (Baseline); n=499 | 2.4 (0.9)
  Change from Baseline to Visit 3 (6 Months); n=450 | 0.2 (0.8)
  Change from Baseline to Visit 5 (12 months); n=406 | 0.4 (0.9)

17. Secondary Outcome: Change From Baseline in Urea Levels at Months 6 and 12
Description: The urea normal range was 10-50 mg/dL.
Time Frame: Baseline, Month 6, Month 12
Population: All participants. n=number of participants with evaluable data at given time-points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
mg/dL
  Before Study Treatment (Baseline); n=494 | 99.0 (40.3)
  Change from Baseline to Visit 3 (6 Months); n=443 | 2.2 (32.1)
  Change from Baseline to Visit 5 (12 months); n=399 | 7.2 (35.3)

18. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (ALP) Levels at Months 6 and 12
Description: The alkaline phosphatase normal range was 40-129 IU/L.
Time Frame: Baseline, Month 6, Month 12
Population: All participants. n=number of participants with evaluable data at given time-points.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
IU/L
  Before Study Treatment (Baseline); n=329 | 124.0 (73.4)
  Change from Baseline to Visit 3 (6 Months); n=245 | -5.0 (49.3)
  Change from Baseline to Visit 5 (12 months); n=215 | -10.3 (62.4)

19. Secondary Outcome: Change From Enrollment in Total Cholesterol Levels at Months 6 and 12
Description: The total cholesterol normal range was 130-200 mg/dL.
Time Frame: Enrollment, Month 6, Month 12
Population: All participants. n=number of participants with evaluable data at given time-points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
mg/dL
  Visit 1 (Enrollment); n=367 | 186.3 (43.3)
  Change from Enrollment to Visit 3 (6 Months);n=272 | -3.8 (38.1)
  Change from Enrollment to Visit 5(12 months);n=243 | -5.4 (39.6)

20. Secondary Outcome: Change From Enrollment in Triglyceride Levels at Months 6 and 12
Description: The normal range for triglycerides was 0-200 mg/dL.
Time Frame: Enrollment, Month 6, Month 12
Population: All participants. n=number of participants with evaluable data at given time-points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
mg/dL
  Visit 1 (Enrollment); n=353 | 151.0 (80.5)
  Change from Baseline to Visit 3 (6 Months); n=259 | -10.2 (56.0)
  Change from Baseline to Visit 5 (12 months); n=228 | -10.3 (64.5)

21. Secondary Outcome: Change From Enrollment in Low Density Lipoprotein Cholesterol (LDL-C) Levels at Months 6 and 12
Description: The LDL-C normal range was 0-150 mg/dL.
Time Frame: Enrollment, Month 6, Month 12
Population: All participants. n=number of participants with evaluable data at given time-points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
mg/dL
  Visit 1 (Enrollment); n=234 | 106.8 (42.8)
  Change from Baseline to Visit 3 (6 Months); n=144 | -1.6 (36.2)
  Change from Baseline to Visit 5 (12 months); n=123 | 0.1 (48.3)

22. Secondary Outcome: Change From Enrollment in High Density Lipoprotein Cholesterol (HDL-C) Levels at Months 6 and 12
Description: The HDL-C normal range was 35-90 mg/dL.
Time Frame: Enrollment, Month 6, Month 12
Population: All participants. n=number of participants with evaluable data at given time-points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
mg/dL
  Enrollment (Visit 1); n=271 | 49.8 (16.6)
  Change from Baseline to Visit 3 (6 Months); n=193 | -1.1 (18.7)
  Change from Baseline to Visit 5 (12 Months); n=166 | -0.7 (20.2)

23. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) Levels at Months 6 and 12
Description: The CRP normal range was 0-0.6 mg/dL.
Time Frame: Baseline, Month 6, Month 12
Population: All participants. n=number of participants with evaluable data at given time-points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
mg/dL
  Before Study Treatment (Baseline); n=149 | 1.9 (3.3)
  Change from Baseline to Visit 3 (6 Months); n=110 | -0.8 (2.6)
  Change from Baseline to Visit 5 (12 Months); n=101 | 0.5 (4.5)

24. Secondary Outcome: Homocysteine Values Throughout the Study
Description: The homocysteine normal range 3.5-20 μmol/L.
Time Frame: Baseline, Enrollment Visit, Month 6, Month 12
Population: All participants. n=the number of participants with evaluable data at given time-points.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Number analyzed (Participants) | 500
μmol/L
  Before Study Treatment (Baseline); n=16 | 24.8 (6.9)
  Visit 1 (Enrollment); n=52 | 24.3 (9.5)
  Visit 2 (3 Months Post-Enrollment); n=35 | 23.2 (7.5)
  Visit 3 (6 Months Post-Enrollment); n=15 | 23.4 (8.2)
  Visit 4 (9 Months Post-Enrollment); n=17 | 24.7 (8.0)
  Visit 5 (12 Months Post-Enrollment); n=13 | 22.4 (10.1)

ADVERSE EVENTS:
Time Frame: All adverse events were collected during the study up to 12 months. Serious adverse events were collected up to 30 days after the end of study.
Arm/Group | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism
Serious Adverse Events (participants affected / at risk) | 19/500
Other Adverse Events (participants affected / at risk) | 168/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism (N=500)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Pyrexia (General disorders) | 3
Asthenia (General disorders) | 1
Oedema peripheral (General disorders) | 1
Ulcer (General disorders) | 1
Unevaluable event (General disorders) | 1
Pneumonia (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Renal failure chronic (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Fluid intake reduced (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Stent placement (Surgical and medical procedures) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Extrapyramidal disorder (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Cerebral microangiopathy (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Kidney Disease (CKD), Secondary Hyperpathyroidism (N=500)
Chronic Kidney Failure (Renal and urinary disorders) | 168

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.